CLINICAL TRIAL: NCT05998759
Title: A Randomized, Double-blind Placebo-controlled Study of Recombinant Human B Lymphocyte Stimulating Factor Receptor-Fc Fusion Protein for the Treatment of Connective Tissue Disease-associated Thrombocytopenia
Brief Title: Telitacicept for the Treatment of Connective Tissue Disease-associated Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of China University of Science and Technology (Anhui Provincial) (Other); Peking University People's Hospital (Other); Peking University Third Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Second Xiangya Hospital of Central South University (Other); Xiangya Hospital of Central South University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); First Hospital of China Medical University (Other); Shandong Provincial Hospital (Other Government); Changhai Hospital (Other); RenJi Hospital (Other); Shanxi Bethune Hospital (Other); West China Hospital (Other); Institute of Hematology & Blood Diseases Hospital, China (Other); Tianjin First Central Hospital (Other); Tianjin Medical University General Hospital (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); The First People's Hospital of Yunnan (Other)
Responsible Party: Principal Investigator, Yongjing Cheng, Professor, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BJ-2021-235; BJ-2021-235 (Other Grant/Funding Number: National High Level Hospital Clinical Research Funding); RCTAIIRCTD001 (Other Grant/Funding Number: RemeGen Go., Ltd)
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Connective Tissue Diseases; Thrombocytopenia
Keywords: Connective Tissue Diseases; Thrombocytopenia; biological agents; B cell; targeted therapy
MeSH Terms: conditions — Connective Tissue Diseases; Thrombocytopenia | interventions — telitacicept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telitacicept plus standard therapy (Experimental): Telitacicept (160mg ih qw for 24 weeks) combined with standard therapy. Standard therapy refers to the following treatment (monotherapy or in combination): glucocorticoid, hydroxychloroquine, and other immunosuppressants (i.e. cyclophosphamide, cyclosporine, mycophenolate mofetil, azathioprine, tacrolimus, methotrexate and leflunomide, et al.).
  Interventions: Biological: Telitacicept
- Placebo plus standard therapy (Placebo Comparator): Placebo combined with standard therapy. Standard therapy refers to the following treatment (monotherapy or in combination): glucocorticoid, hydroxychloroquine, and other immunosuppressants (i.e. cyclophosphamide, cyclosporine, mycophenolate mofetil, azathioprine, tacrolimus, methotrexate and leflunomide, et al.).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Telitacicept — subcutaneous telitacicept 160 mg weekly for 24 weeks.
  Other Names: recombinant human B lymphocyte stimulating factor receptor-Fc fusion protein; Recombinant Human B Lymphocyte(RC18); Tai'ai®
  Arms: Telitacicept plus standard therapy
Drug: Placebo — subcutaneous placebo weekly for 24 weeks.
  Other Names: Placebo control; control
  Arms: Placebo plus standard therapy

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Telitacicept for the treatment of connective tissue disease-associated thrombocytopenia.

DETAILED DESCRIPTION:
In this randomized, double-blind placebo-controlled study, the investigators aim to evaluate the efficacy and safety of Telitacicept for the treatment of connective tissue disease-associated thrombocytopenia. After screening, eligible participants will be randomized at a 1: 1 ratio to receive either subcutaneous Telitacicept 160 mg or placebo once a week for 24 weeks. The background standard therapy is maintained stable during the whole treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been diagnosed with connective tissue disease (CTD)-associated thrombocytopenia. And CTD includes primary Sjögren syndrome (according to the 2002 American College of Rheumatology (ACR)/ European League against Rheumatism (EULAR) classification criteria), systemic lupus erythematosus (SLE, according to the 1997 or the 2009 ACR classification criteria), and undifferentiated connective tissue disease (according to the 1999 international classification criteria)
* Refractory thrombocytopenia defined as:

Either: Failure to maintain sustained remission after treatment by glucocorticoid and at least one immunosuppressant (i.e. cyclophosphamide, cyclosporine, mycophenolate mofetil, azathioprine, tacrolimus, methotrexate, leflunomide and hydroxychloroquine, et al.) Or: Relapse during oral glucocorticoid tapering or after withdrawal

* 50×10^9/L>PLT
* anti-nuclear antibody (ANA) positive (≥1:80, any karyotype) detected in the laboratory of each research center
* Standard therapy should be maintained stable for at least 14 days prior to the first dose of the experimental drug or placebo. Standard therapy refers to the following treatment (monotherapy or in combination): glucocorticoid, hydroxychloroquine, and other immunosuppressants (i.e. cyclophosphamide, cyclosporine, mycophenolate mofetil, azathioprine, tacrolimus, methotrexate and leflunomide, et al.)
* Signed informed consent form, willing or able to participate in all required study evaluations and procedures

Exclusion Criteria:

* Vital organ lethal bleeding (including but not limited to central nervous system bleeding, digestive tract bleeding) at screening, or intracranial bleeding 6 months prior to screening
* Antiphospholipid syndrome, thrombotic thrombocytopenia purpura, hemolytic uremic syndrome, or thrombocytopenia secondary to other causes (such as sepsis, Epstein-Barr virus infection, cytomegalovirus infection, Corona Virus Disease-19 (COVID-19) infection, drugs, etc.)
* Hematopoietic system disorders, such as myelodysplastic syndrome, paroxysmal sleep hemoglobinuria, aplastic anemia, leukemia, lymphoma, myelofibrosis and so on
* Severe cardiovascular system disease, including: unstable or uncontrollable disease or condition affecting the function of the heart (such as angina pectoris, congestive heart failure, uncontrolled hypertension or arrhythmia)
* Arteriovenous thromboembolism events
* Receiving antiplatelet or anticoagulant therapy at screening
* Clinically significant electrocardiogram changes
* corrected Q-T interval (QTc)>450ms for male, QTc>470ms for female
* Severe pulmonary disease, including: unstable or uncontrollable disease or condition affecting respiratory function [e.g., diffuse alveolar hemorrhage, severe pulmonary hypertension, severe pulmonary interstitial disease (peripheral blood oxygen saturation <92% at rest without oxygen, or forced vital capacity (FVC)<50%, or carbon monoxide diffusing capacity (DLCO)<50%)]
* Severe kidney disease, including: severe lupus nephritis (urinary protein > 6 g/24 hours or endogenous creatinine clearance < 30 ml /min) 8 weeks prior to randomization, active nephritis requiring current protocol disallowed drugs, severe renal insufficiency requiring hemodialysis or prednisone ≥100mg/ day (or equivalent) for ≥14 days
* SLE or non-SLE related central nervous system disease (including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident, encephalitis, central nervous system vasculitis) 8 weeks prior to randomization
* Active hepatitis, a history of severe liver disease. Subjects positive for hepatitis B surface antigen (HBsAg) or antibodies to hepatitis C virus are excluded. As for subjects with antibodies to hepatitis B core antigen (HBcAb), further hepatitis B virus (HBV)-DNA should be tested. If HBV-DNA is negative, subjects could be enrolled; otherwise, subjects should be excluded
* Abnormal laboratory results (including but not limited to: alanine aminotransferase (ALT) or aspertate aminotransferase (AST)≥3×ULN (upper limit of normal), white blood cell count <1.5×10^9/L)
* Subjects with known active infections (e.g., shingles, COVID-19, HIV, active tuberculosis, etc.), and active or recurrent gastrointestinal ulcers
* Pregnant or lactating women, and subjects with a during plan during the trial
* Allergic reaction: history of allergic reactions to human biological products
* Treatment with B cell-targeting agents such as Rituximab or Epratuzumab or Belimumab six months prior to randomization
* Treatment with tumor necrosis factor (TNF) inhibitors or TNF-receptor blockers six months prior to randomization
* Participating in clinical trial 28 days or 5 drug half-lives of the investigational agents prior to randomization
* Received live vaccine 28 days prior to randomization
* Treatment with unstable dosage of thrombopoietin receptor agonists such as Eltrombopag or Romiplostim 14 days prior to randomization
* Subjects with depression or suicidal thoughts
* Previous treatment with telitacicept
* B cell targeting drug therapy is not tolerated or responsive
* Investigator considers candidates not appropriating for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2023-12-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall response (CR + PR) rate | at week 24
  Response is deemed as complete (CR) if the platelet (PLT) count is ≥ 100×10^9/L, partial (PR) if the platelet count ranges from 50×10^9/L to 100×10^9/L and at least doubled from baseline. No active bleeding is allowed in participants classified as CR or PR.

SECONDARY OUTCOMES:
Overall response (CR + PR) rate | at week 12
  Response is deemed as complete (CR) if the platelet count is ≥ 100×10^9/L, partial (PR) if the platelet count ranges from 50×10^9/L to 100×10^9/L and at least doubled from baseline. No active bleeding is allowed in participants classified as CR or PR.
Rescue treatment rate | at week 24
  Rescue treatment is initiated if the platelet count is <10×10^9/L, or the participant is with active bleeding, or based on the investigator's judgement when the platelet count ranges from 10×10^9/L to 30×10^9/L.
Time to rescue treatment | at week 24
  Time to rescue treatment refers to period duration from the initiation of Telitacicept or placebo (day 1) to rescue treatment.
Relapse rate | at week 24
  No response refers to the platelet count is < 50×10^9/L, or increases for less than 1-fold from baseline, or with active central nervous system or digestive tract bleeding, or rescue treatment is initiated. Relapse is defined as no response recurring after a complete or partial response lasting for at least 7 days with treatment.
Time to relapse | at week 24
  Time to relapse refers to period duration from the initiation of Telitacicept or placebo (day 1) to relapse.
treatment related adverse event | at week 24
  According to the NCI CTCAE 5.0
treatment related severe adverse event | at week 24
  According to the NCI CTCAE 5.0
bleeding scale | at week 24
  According to the ITP bleeding scale (IBLS). The IBLS comprises of 11 grades from 0 (none) to 2 (marked bleeding) by history over the previous week or by exam; 2 being worse. These 11 grades include: skin by physical exam, oral by physical exam, skin by history, oral by history, epistaxis, gastrointestinal, urinary, gynecological, pulmonary, intracranial hemorrhage, and subconjunctival hemorrhage.

OTHER OUTCOMES:
life quality 1 | at week 24
  According to the ITP Patient Assessment Questionnaire™ (ITP-PAQ™) score. The ITP-PAQ™ is a disease-specific instrument that was designed to measure the Quality of Life (QoL) of adult patients with immune thrombocytopenia. The items employ a 4-week recall with responses recorded on 4-, 5- or 7-point Likert scales. All item scores are transformed to a 0 to 100 continuum where higher scores represent better QoL and are weighted equally to derive the scale scores.
life quality 2 | at week 24
  According to the FACT-Th6 score. The Functional Assessment of Cancer Therapy-Thrombocytopenia (FACT-Th6) consists of 6 questions in which patients rate (0-4) their general degree of worry related to bleeding and bruising, and resulting activity impairment and frustration. Items were reverse-scored as necessary such that higher scores represent higher Health-related quality of life (HRQoL). Total scores ranged from 0 to 24. Recall period is previous 7 days.
Absolute change rate from baseline in serum immunoglobulin G (IgG) | at week 24
  (serum IgG level at week 24-serum IgG level at baseline)/ serum IgG level at baseline
Absolute change rate from baseline in serum immunoglobulin M (IgM) | at week 24
  (serum IgM level at week 24-serum IgM level at baseline)/ serum IgM level at baseline
Absolute change rate from baseline in serum immunoglobulin A (IgA) | at week 24
  (serum IgA level at week 24-serum IgA level at baseline)/ serum IgA level at baseline
Absolute change rate from baseline in serum C3 | at week 24
  (serum C3 level at week 24-serum C3 level at baseline)/ serum C3 level at baseline
Absolute change rate from baseline in serum C4 | at week 24
  (serum C4 level at week 24-serum C4 level at baseline)/ serum C4 level at baseline
Absolute change rate from baseline in serum anti-platelet antibody | at week 24
  (serum anti-platelet antibody level at week 24-serum anti-platelet antibody level at baseline)/ serum anti-platelet antibody level at baseline
Absolute change rate from baseline in serum Blys | at week 24
  (serum Blys level at week 24-serum Blys level at baseline)/ serum Blys level at baseline. Blys is short for B lymphocyte stimulator.
Absolute change rate from baseline in serum APRIL | at week 24
  (serum APRIL level at week 24-serum APRIL level at baseline)/ serum APRIL level at baseline. APRIL is short for a proliferation-inducing ligand.
Absolute change rate from baseline in peripheral naive B cell count | at week 24
  (peripheral naive B cell count at week 24-peripheral naive B cell count at baseline)/ peripheral naive B cell count at baseline.
Absolute change rate from baseline in peripheral plasma cell count | at week 24
  (peripheral plasma cell count at week 24-peripheral plasma cell count at baseline)/ peripheral plasma cell count at baseline.
Absolute change rate from baseline in peripheral plasmablast count | at week 24
  (peripheral plasmablast count at week 24-peripheral plasmablast count at baseline)/ peripheral plasmablast count at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Zhang, MD., Study Chair — Beijing Hospital; Yongjing Cheng, MD., Study Chair — Beijing Hospital; Shengqian Xu, MD., Principal Investigator — The First Affiliated Hospital of Anhui Medical Hospital; Zhu Chen, MD., Principal Investigator — The First Affiliated Hospital of China University of Science and Technology (Anhui Provincial); Jing He, MD., Principal Investigator — Peking University People's Hospital; Rong Mu, MD., Principal Investigator — Peking University Third Hospital; Niansheng Yang, MD., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Yang Li, MD., Principal Investigator — Guangdong Provincial People's Hospital; Guanmin Gao, MD., Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Anbin Huang, MD., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Fen Li, MD., Principal Investigator — Second Xiangya Hospital of Central South University; Hui Luo, MD., Principal Investigator — Xiangya Hospital of Central South University; Hongbin Li, MD., Principal Investigator — The Affiliated Hospital of Inner Mongolia Medical University; Pinting Yang, MD., Principal Investigator — First Hospital of China Medical University; Hongsheng Sun, MD., Principal Investigator — Shandong Provincial Hospital; Dongbao Zhao, MD., Principal Investigator — Changhai Hospital; Sheng Chen, MD., Principal Investigator — RenJi Hospital; Liyun Zhang, MD., Principal Investigator — Shanxi Bethune Hospital; Qibing Xie, MD., Principal Investigator — West China Hospital; Lei Zhang, MD., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China; Wufang Qi, MD., Principal Investigator — Tianjin First Central Hospital; Wei Wei, MD., Principal Investigator — Tianjin Medical University General Hospital; Lijun Wu, MD., Principal Investigator — People's Hospital of Xinjiang Uygur Autonomous Region; Qin Li, MD., Principal Investigator — The First People's Hospital of Yunnan
Locations (23):
- China (23):
  - The First Affiliated Hospital of Anhui Medical College, Hefei, Anhui
  - The First Affiliated Hospital of China University of Science and Technology (Anhui Provincial), Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital, China, Wuhan, Hubei
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - RenJi Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang Uygur Autonomous Region
  - The First People's Hospital of Yunnan, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No